CLINICAL TRIAL: NCT02138773
Title: A Randomized, Single Dose, Open-label, Cross-over Study on Bioequivalence of Two Formulations of Tamsulosin Hydrochloride Prolonged Release Capsule (Tamsulosin Pellet From Meppel Plant and Nishine Plant) Under Fed and Fasted Conditions in Chinese Healthy Male Subjects
Brief Title: A Study to Compare How Tamsulosin is Absorbed to the Body After Administration of Two Types of Tamsulosin Formulation Under Fed and Fasted Conditions in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 617-CL-CN3
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Healthy; Pharmacokinetics of Tamsulosin Hydrochloride
Keywords: prolonged release formulation; adrenergic blocker; Bioequivalence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fed, formulation-A (Experimental): drug administered at 0.5h after the start of a standard breakfast
  Interventions: Drug: Tamsulosin formulation-A
- Fed, formulation-B (Experimental): drug administered at 0.5h after the start of a standard breakfast
  Interventions: Drug: Tamsulosin formulation-B
- Fasted, formulation-A (Experimental): drug administered under fasted condition (fasting for at least 10 hours)
  Interventions: Drug: Tamsulosin formulation-A
- Fasted, formulation-B (Experimental): drug administered under fasted condition (fasting for at least 10 hours)
  Interventions: Drug: Tamsulosin formulation-B

INTERVENTIONS:
Drug: Tamsulosin formulation-A — oral
  Other Names: Harnal
  Arms: Fasted, formulation-A; Fed, formulation-A
Drug: Tamsulosin formulation-B — oral
  Other Names: Harnal
  Arms: Fasted, formulation-B; Fed, formulation-B

SUMMARY:
The purpose of this study is to investigate the relative bioavailability of two types of prolonged release formulation of tamsulosin hydrochloride in Chinese healthy subjects. The safety of tamsulosin formulation is also compared.

DETAILED DESCRIPTION:
There will be two studies. One study will be conducted under fed condition, and the other study will be conducted under fasted condition. Each study is a single center, randomized, single dose, open-labeled, cross-over study.

Study 1 will be conducted under fed condition:

Subjects will undergo screening evaluations to determine their eligibility within 7 days prior to the study enrollment. Subjects will be admitted to the clinical facility in the evening prior to dosing for each period. All subjects will receive tamsulosin formulation-A and formulation-B in one of two randomly assigned treatment sequences at 0.5h after the start of a standard breakfast. There will be a 7-day washout period between each dose.

Study 2 will be under fasted condition:

A single oral dose of tamsulosin formulation-A or formulation-B will be given to subjects under fasted condition (fasting for at least 10 hours since 20:00PM the night before the administration). Blood will be sampled at the same time point as in Study 1. Also, safety evaluation will be performed at the same selected times throughout the study as in Study 1.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI=weight (kg)/height(m)2) between 19 and 24 (included)
* Body weight no less than 50 kg
* Healthy as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs and clinical laboratory determinations

Exclusion Criteria:

* Subject receiving drug treatment (including OTC) within 4 weeks prior to the first administration
* Subject with a known or suspected history of allergic condition and/or hypersensitivity to Tamsulosin, any excipients in the drug product or drugs of the same class
* Existing cardiac, haematological, hepatic, renal, gastrointestinal or any other acute or chronic disease and/or pathological findings, which might interfere with the drug's safety, tolerability, absorption and/or pharmacokinetics
* Subject with symptomatic hypotension whatever the decrease of blood pressure or asymptomatic postural hypotension defined by a decrease in SBP or DBP equal to or greater than 20mmHg within two minutes when changing from the supine to the standing position
* Subject with sitting DBP<60mmHg or >90mmHg, and/or SBP<90mmHg or>140mmHg, and/or pulse rate (PR) <40/min or >90/min, and/or axilla temperature >37℃ or <35℃ within the screen period
* Subject with a previous history of drug abuse or subject showing any degree of drug abuse within 3 months prior to the present study
* Subject with a blood donation or other plasma loss of more than 200mL or received a transfusion of any blood or blood products within 3 months prior to the start of the present study
* Subject with a treatment of plasma exchange within 4 weeks prior to the present study
* Subject participated in any other study within 3 months prior to the present study, or participated in more than 3 studies during the last 12 months prior to the start of the present study
* Subject with HBs-Ag, HCV-Ab or HIV-Ab
* Subject with a partner wish to become pregnant during the present study period and 30 days after the study
* Subject is mentally or physically disabled

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of tamsulosin (AUC0-t) | up to 72 hr after administration
  AUC0-t will be calculated according to the linear trapezoidal rule.
Pharmacokinetic parameter of tamsulosin (Cmax) | up to 72 hr after administration

SECONDARY OUTCOMES:
Pharmacokinetic parameter of tamsulosin (AUC0-∞) | up to 72 hr after administration
Pharmacokinetic parameter of tamsulosin (Tmax) | up to 72 hr after administration
Pharmacokinetic parameter of tamsulosin (T1/2) | up to 72 hr after administration
Safety evaluated by physical examinations, vital signs, electrocardiograms, laboratory assessments, and adverse events. | up to 72 hr after administration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Shanghai, China